CLINICAL TRIAL: NCT03929003
Title: Breathe Free: Smartphone Videogame-Based Incentives for Smoking Cessation
Brief Title: Inspired: Smartphone Videogame-Based Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProG0520140170
Record Dates: First submitted 2017-09-26; First posted 2019-04-26 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: Two group randomization
Who Masked: Participant
Masking Description: Participants will not be told whether they are in the control or experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingent (Experimental): Participants in this arm will be required to meet CO goals in order to earn game-based rewards.
  Interventions: Behavioral: Inspired
- Non-contingent (Active Comparator): Participants in this arm will submit CO verifications but will earn game-based rewards independent of meeting CO goals.
  Interventions: Behavioral: Inspired

INTERVENTIONS:
Behavioral: Inspired — The investigators will be studying the ability of using videogame-based rewards to increase smoking abstinence when they are made contingent on meeting abstinence goals.

SUMMARY:
The investigators are testing a new, smartphone videogame-based intervention for smoking cessation.

DETAILED DESCRIPTION:
The investigators have developed a novel smartphone videogame, where smokers are required to submit breath carbon monoxide samples to demonstrate smoking abstinence, and where they will earn game-based rewards contingent on meeting CO goals. Players will be working with teams to earn group and social rewards to help advance their game.

ELIGIBILITY:
Inclusion Criteria:

* Inclusionary criteria: Participants will be required to be of legal smoking age (>19 in Alabama, Alaska, New Jersey, Utah, and in Onondaga, Nassau and Suffolk Counties in New York, > 18 years of age in the remainder of the United States). Participants must also report smoking >10 cigarettes per day, report smoking for >2 years, answer 8 or higher on a Likert scale asking how much the person wishes to quit smoking right now (1 = not at all, 10 =very much), have a smartphone with a data plan and active contract extending for at least two months from the enrollment date (i.e., the duration of the study), and reside in the U.S. Participants in the study must submit an initial CO reading > 10ppm (to prevent nonsmokers from enrolling in the study), Literacy will be assessed by having the participant read the first few lines of the consent form out loud, and will be an inclusion criterion because elements of "Breathe Free" will require reading.

Exclusion Criteria:

* Individuals will be excluded from the study if they report smoking any combustible products >2 times per month, report unstable medical/psychiatric conditions that might interfere with the study objectives (e.g., asthma), report living with someone who smokes in the house, or has a career that results in excessive exposure to CO. All excluded participants will be emailed the following smoking cessation information: the "Clearing the Air" packet developed by the National Cancer Institute, Smokefree.gov, Quitsmokinghelpline.com, and the National Academies Press "Dying to quit."

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 7 days
  self-report of smoking abstinence over the previous 7-day period.

SECONDARY OUTCOMES:
Demographic | 7 weeks
  description of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodwin S, Nastasi JA, Newman ST, Rapoza D, Raiff BR. Feasibility and Acceptability of a Mobile Game to Support Smoking Cessation: Repeated Measures Study. JMIR Serious Games. 2024 Aug 21;12:e54684. doi: 10.2196/54684. PMID 39167443
- [Derived] Upton CR, Nastasi JA, Raiff BR. Identifying Video Game Preferences Among Adults Interested in Quitting Smoking Cigarettes: Survey Study. JMIR Serious Games. 2022 Mar 24;10(1):e30949. doi: 10.2196/30949. PMID 35323116